CLINICAL TRIAL: NCT05706805
Title: NAVISCORE Post-Market Clinical Follow-up Study
Brief Title: NAVISCORE PMCF Study ( rEPIC04F )
Acronym: rEPIC04F
Status: Completed | Type: Observational
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Other Study IDs: NAVISCORE PMCF Study
Record Dates: First submitted 2022-11-15; First posted 2023-01-31 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Coronary Artery Disease; Ischemic Heart Disease
Keywords: MDR (Medical Device Regulations); PMCF (Post-Market Clinical Follow-up); Coronary balloon dilatation catheter
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary Artery Disease (CAD)
  Interventions: Device: Naviscore

INTERVENTIONS:
Device: Naviscore — Patients in whom treatment with (Naviscore) has been attempted

SUMMARY:
Multicenter, prospective, non-randomized, post-market clinical follow-up (PMCF) study to confirm and support the clinical safety and performance of Naviscore scoring balloon to meet EU Medical Device regulation (MDR) requirements in all the CONSECUTIVE patients treated with Naviscore.

DETAILED DESCRIPTION:
The objective of this multicenter, prospective, non-randomized, post-market clinical follow-up (PMCF) study is to confirm and support the clinical safety and performance of the Naviscore scoring balloon in a NON-SELECTED, Real World population under daily clinical practice when used as intended by the manufacturer to meet EU Medical Device regulation requirements for post-market clinical follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient treated with Naviscore according to routine hospital practice and following instructions for use
* Informed consent signed

Exclusion Criteria:

• Not meet inclusion criteria

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients treated with Naviscore according to routine hospital practice and following instructions for use
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
Safety Endpoint. Freedom from Target Lesion Failure | 7 days
  Freedom from TARGET LESION FAILURE (TLF), composite endpoint of cardiac death, myocardial infarction (MI) and a new Target Lesion Revascularization (TLR).

SECONDARY OUTCOMES:
Efficacy Endpoint. Freedom from Target Lesion Failure (TLF) | 7 days
  Freedom from TARGET LESION FAILURE (TLF), composite endpoint of Cardiac death, Myocardial infarction, and new Target Lesion Revascularization (TLR).
Freedom from Balloon rupture | During PCI (Percutaneous Coronary Intervention)
  Freedom from Balloon rupture
Freedom from Hypotube rupture | During PCI (Percutaneous Coronary Intervention)
  Freedom from Hypotube rupture ( partial or total fracture of the shaft of the device)
Freedom from Complicated withdrawal | During PCI (Percutaneous Coronary Intervention)
  Freedom from Complicated withdrawal (difficult or impossible device retrieval that may or may not cause clinical complications)
Freedom from Coronary perforation | During PCI (Percutaneous Coronary Intervention)
  Freedom from Coronary perforation according to the modified Ellis classification
Freedom from Coronary dissection >C | During PCI (Percutaneous Coronary Intervention)
  Freedom from Coronary dissection >C according to the NHLBI Classification (National Heart, Lung, and Blood Institute)
Freedom from No reflow | During PCI (Percutaneous Coronary Intervention)
  Freedom from No reflow (persistently slowed flow with residual stenosis <30% and no flow-limiting dissection)
Freedom from Coronary thrombosis | During PCI (Percutaneous Coronary Intervention)
  Freedom from Coronary thrombosis according to ARC-2 ( Academic Research Consortium-2) criteria

CONTACTS AND LOCATIONS:
Locations (7):
- Spain (7):
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario de Cáceres, Cáceres
  - Hospital Universitario Juan Ramon Jimenez, Huelva
  - Hospital Universitario de Leon, León
  - Hospital Universitario Lucus Agusti, Lugo
  - Hospital Regional Universitario Carlos Haya, Málaga

REFERENCES:
- [Background] Fonseca A, Costa Jde R Jr, Abizaid A, Feres F, Abizaid AS, Costa R, Staico R, Mattos LA, Sousa AG, Grube E, Sousa JE. Intravascular ultrasound assessment of the novel AngioSculpt scoring balloon catheter for the treatment of complex coronary lesions. J Invasive Cardiol. 2008 Jan;20(1):21-7. PMID 18174614
- [Background] Weisz G, Metzger DC, Liberman HA, O'Shaughnessy CD, Douglas JS Jr, Turco MA, Mehran R, Gershony G, Leon MB, Moses JW. A provisional strategy for treating true bifurcation lesions employing a scoring balloon for the side branch: final results of the AGILITY trial. Catheter Cardiovasc Interv. 2013 Sep 1;82(3):352-9. doi: 10.1002/ccd.24630. Epub 2013 Mar 9. PMID 22927100
- [Background] US FDA: Summary of Safety and Effectiveness Data (SSED): AngioSculpt®Scoring Balloon Catheter (2007) www.accessdata.fda.gov/cdrh_docs/pdf5/P050018b.pdf